Accuracy of computer-assisted template-based implant placement using CAD/CAM stereolithographic surgical templates with or without metallic sleeves: a randomized controlled trial

Marco Tallarico

### Randomization

One computer-generated restricted randomization list was created. Only one of the investigators, not involved in the selection and treatment of the patients, was aware of the random sequence and could have access to the randomization lists stored in a password-protected portable computer. The random codes were enclosed in sequentially numbered, identical, opaque, sealed envelopes. Envelopes were opened sequentially after the prosthetic-driven plan was approved.

## Statistical analysis

Patient data were collected in a Numbers spreadsheet (Version 3.6.1 for Mac OS X 10.11.4). A bio-statistician with expertise in dentistry analyzed the data using SPSS software for Mac OS X (version 22.0; SPSS Inc., Chicago, IL, USA) for statistical analysis. Descriptive analysis was performed for numeric parameters using mean±standard deviation and median with confidence interval (95% CI). Implant failure and template-related complications between the two groups were compared using Fisher's exact probability test. The mean differences of the overall deviation in the clinical outcomes compared to the virtual plan, were compared between groups using a mixed-model repeated-measures analysis of variance (ANOVA). In the sleeve-less group, accuracy of open versus closed holes were also evaluated. All statistical comparisons were conducted with a P value set at 0.05.

### **Results**

Thirty-two patients were considered eligible for this trial. Two patient was not included due to them not wanting to participate in this study. No patient dropped out, and all patients were treated according to the allocated interventions.

Fifteen patients (8 female and 7 male with a mean age of 45.1 years) were randomised to the control group (template with metallic sleeves) and 15 (10 female and 5 male with a mean age of 55.2 years) to the test group (without metallic sleeves). A total of 37 implants were placed in the control group while 43 implants were placed in the test group. Of these, 12 implants were placed through open sleeves and 31 through closed sleeves.

No implants failed and no complications were experienced. All the implants were inserted according to the manufacturer's instructions, with an insertion torque ranged between 35 an 45 Ncm.

In the control group, the analysis of the final implant accuracy revealed a total mean error of 2.25±1.41° (range 0.3–5.0°; 95% CI 0.52 to 1.65°) in angle; 0.52±0.30 mm (range 0.1–1.1 mm; 95% CI 0.39 to 0.61 mm) in the horizontal plan (mesio-distal), and 0.58±0.44 mm (range 0.0–1.6 mm; 95% CI 0.44 to 0.76 mm) in the vertical plan (apico-coronal).

Overall, in the test group, the analysis of the final implant accuracy revealed a total mean error of 1.61±1.90° (range 0.1–6.8°; 95% CI 0.17 to 1.31°) in angle; 0.54±0.41 mm (range 0.05–1.7 mm; 95% CI 0.31 to 0.55 mm) in the horizontal plan (mesio-distal), and 0.37±0.27 mm (range 0.0–1.3 mm; 95% CI 0.23 to 0.39 mm) in the vertical plan (apico-coronal).

Sub group analysis relieved a mean error in angle of  $2.89\pm2.36^{\circ}$  (range  $0.2-6.8^{\circ}$ ; 95% CI 1.41 to  $4.09^{\circ}$ ) with open sleeves and  $1.20\pm1.43^{\circ}$  (range  $0.1-5.9^{\circ}$ ; 95% CI 0.2 to  $1.2^{\circ}$ ) with closed sleeves; the differences was statistically significant (P = 0.0357). In the horizontal plan (mesio-distal), the mean error was  $0.73\pm0.49$  mm (range 0.2-1.5 mm; 95% CI 0.37 to 0.93 mm) with open sleeves and  $0.49\pm0.38$  mm (range 0.05-1.7 mm; 95% CI 0.27 to 0.53 mm) with closed sleeves; the

difference was not statistically significant (P = 0.1553). In the vertical plan (apico-coronal), the mean error was  $0.43\pm0.34$  mm (range 0.0-1.0 mm; 95% CI 0.16 to  $0.54^{\circ}$ ) with open sleeves and  $0.33\pm0.25$  mm (range 0.05-1.3 mm; 95% CI 0.21 to 0.39 mm) with closed sleeves; the difference was not statistically significant (P = 0.4048).

Comparing the mean value of the control group (closed metallic sleeves) with mean value of the closed sleeves of the test group. There was a statistically significant difference in angle (P = 0.0063) and in the vertical plan (P = 0.0126) with lower values in the test group. While, there was not statistically significant difference in the horizontal plan (P = 0.7546).

**Conclusions:** With the limitation of the present randomized controlled trial, intraoral digital impression may be a viable option for the rehabilitation of partial edentulous patients when computerguided template-assisted implant placement is used. Furthermore, intraoral digital impression reduces the number of appointments, resulting in shorter treatment time. In both groups, the maximum tridimensional deviations (angular, horizontal, vertical) did not exceed the safe offset of the software.

### References

Ahlholm, P., Sipila, K., Vallittu, P., Jakonen, M. & Kotiranta, U. (2016) Digital Versus Conventional Impressions in Fixed Prosthodontics: *A Review. Journal of Prosthodontics* Aug 2. doi: 10.1111/jopr.12527. [Epub ahead of print]

Canullo, L., Tallarico, M., Radovanovic, S., Delibasic, B., Covani, U. & Rakic, M. (2016) Distinguishing predictive profiles for patient-based risk assessment and diagnostics of plaque induced, surgically and prosthetically triggered peri-implantitis. *Clinical Oral Implants Research* 27: 1243–50.

Chochlidakis, K.M., Papaspyridakos, P., Geminiani, A., Chen, C.-J., Feng, I.J. & Ercoli, C. (2016) Digital versus conventional impressions for fixed prosthodontics: A systematic review and meta-analysis. *The Journal of Prosthetic Dentistry* **116**: 184–190.

D'haese, J., Van De Velde, T., Komiyama, A., Hultin, M. & De Bruyn, H. (2012) Accuracy and complications using computer designed stereolithographic surgical guides for oral rehabilitation by means of dental implants: a review of the literature. *Clinical Implant Dentistry and Related Research* 14: 321–335.

Furhauser, R., Mailath-Pokorny, G., Haas, R., Busenlechner, D., Watzek, G. & Pommer, B. (2015) Esthetics of Flapless Single-Tooth Implants in the Anterior Maxilla Using Guided Surgery: Association of Three-Dimensional Accuracy and Pink Esthetic Score. *Clinical Implant Dentistry and Related Research* 17: e427-433.

Johansson, B., Friberg, B., Nilson, H. (2009) Digitally planned, immediately loaded dental implants with prefabricated prostheses in the reconstruction of edentulous maxillae: a 1-year prospective, multicentre study. *Clinical Implant Dentistry and Related Research* **11**: 194–200.

Jung, R.E., Schneider, D., Ganeles, J., Wismeijer, D., Zwahlen, M., Hämmerle CHF & Tahmaseb, A. (2009) Computer technology applications in surgical implant dentistry: a systematic review. *The International Journal of Oral & Maxillofacial Implants* **24**: 92–109.

Komiyama, A., Klinge, B. & Hultin, M. (2008) Treatment outcome of immediately loaded implants installed in edentulous jaws following computer-assisted virtual treatment planning and flapless surgery. *Clinical Oral Implants Research* **19**: 677–685.

Meloni, SM., De Riu, G., Pisano, M., Cattina, G. & Tullio, A. (2010) <u>Implant treatment software</u> planning and guided flapless surgery with immediate provisional prosthesis delivery in the fully edentulous maxilla. A retrospective analysis of 15 consecutively treated patients. *Eur J Oral Implantol* 3:245-51.

Meloni, SM., De Riu, G., Pisano, M., Lolli, FM., Deledda, A., Campus, G. & Tullio A. (2013a) Implant Restoration of Edentulous Jaws with 3D Software Planning, Guided Surgery, Immediate Loading, and CAD-CAM Full Arch Frameworks. *Int J Dent*. Jul 29.

Meloni, SM., De Riu, G., Pisano, M., Dell'aversana Orabona, G., Piombino, P., Salzano, G., Quarato, D., Riccardi, E., Belli, E. & Ungari, C. (2013b) Computer-assisted implant surgery and immediate loading in edentulous ridges with dental fresh extraction sockets. Two years results of a prospective case series study. *Eur Rev Med Pharmacol Sci.* 17:2968-73.

Meloni, S.M., Tallarico, M., Pisano, M., Xhanari, E. & Canullo, L. (2017) Immediate loading of fixed complete denture prosthesis supported by 4-8 implants placed using guided surgery: a 5 years prospective study on 66 patients with 356 implants. *Clinical Implant Dentistry and Related Research* 19: 195-206.

Merli, M., Bernardelli, F., Esposito, M. (2008) Computer-guided flapless placement of immediately loaded dental implants in the edentulous maxilla. A pilot prospective case series. *European Journal of Oral Implantology* **1**: 61–69.

Polizzi, G., Cantoni, T., Pasini, E. & Tallarico, M. (2016) Immediate loading of variable-thread expanding tapered-body implants placed into maxillary post-extraction or healed sites using a guided surgery approach: An up-to five year retrospective analysis. *Journal of Oral Science & Rehabilitation* 2: 50–60.

Pozzi, A., Tallarico, M., Marchetti, M., Scarfo, B. & Esposito M. (2014) Computer-guided versus free-hand placement of immediately loaded dental implants: 1-year post-loading results of a multicentre randomised controlled trial. *European Journal of Oral Implantology* 7: 229–242.

Tahmaseb, A., Wismeijer, D., Coucke, W. & Derksen W. (2014) Computer technology applications in surgical implant dentistry: a systematic review. *International Journal of Oral & Maxillofacial Implants* **29**: 25–42.

Tallarico, M., Meloni, S.M., Canullo, L., Caneva, M. & Polizzi G. (2016) Five-Year Results of a Randomized Controlled Trial Comparing Patients Rehabilitated with Immediately Loaded Maxillary Cross-Arch Fixed Dental Prosthesis Supported by Four or Six Implants Placed Using Guided Surgery. *Clinical Implant Dentistry and Related Research* **18**: 965-972.

Tallarico, M., Xhanari, E., Cocchi, F., Canullo, L., Schipani, F., & Meloni, S.M. (2017a) Accuracy of computer-assisted template-based implant placement using a conventional impression and scan model or digital impression: A preliminary report from a randomized controlled trial. *Journal of Oral Science & Rehabilitation* **3**: 08–16.

Tallarico, M., & Meloni, S. (2017b) Retrospective Analysis on Survival Rate, Template-Related Complications, and Prevalence of Peri-implantitis of 694 Anodized Implants Placed Using Computer-Guided Surgery: Results Between 1 and 10 Years of Follow-Up. *The International Journal of Oral & Maxillofacial Implants* 32: 1162–1171.

van Steenberghe, D., Glauser, R., Blomback, U., Andersson, M., Schutyser, F., Pettersson, A. & Wendelhag, I. (2005) Computed tomographic scan-derived customized surgical template and fixed prosthesis for flapless surgery and immediate loading of implants in fully edentulous maxillae: a prospective multicentre study. *Clinical Implant Dentistry and Related Research* 2005, 7: 111–120. Vasak, C., Watzak, G., Gahleitner, A., Strbac, G., Schemper, M. & Zechner, W. (2011) Computed tomography-based evaluation of template (NobelGuide<sup>TM</sup>)-guided implant positions: a prospective radiological study. *Clinical Oral Implants Research* 22: 1157–63.

Vermeulen, J. (2016) The Accuracy of Implant Placement by Experienced Surgeons: Guided vs Freehand Approach in a Simulated Plastic Model. *International Journal of Oral & Maxillofacial Implants* **32**: 617–624.

- Figure 1. Virtual implant planning.
- Figure 2. Post-operative STL file derived from the intraoral scan
- Figure 3. Geometrical alignment of the files exported from the planning, and the post-operative STL file by automated image registration.
- Figure 4. The horizontal (lateral), vertical (depth) and angular deviation between virtual and placed implants calculated along the long axis of each implants.
- Figure 5. Maximum angular deviation calculated according to the implant diameter and length.

# Tables

| Table 1. Main patient and implant characteristics. | | | |
|---|---|---|---|
| | Conventional (n=29) | Digital (n=28) | P value |
| Age | 45.4±13 | 43.7±15.7 | 0.795 |
| Female patients | 5 | 6 | 1 |
| Implants placed in the maxilla | 18 | 15 | 0.596 |
| Immediately loaded i plants | 13 | 11 | 0.790 |
| Post-extractive implants | 4 | 1 | 0.352 |
| Sinus lift procedures | 2 | 1 | 1 |
| Complete restorations | 3 | 1 | 0.611 |
| Partial restorations | 3 | 2 | 1 |
| Single restorations | 7 | 18 | 0.003 |

1.